CLINICAL TRIAL: NCT01770912
Title: A Randomized, Double-Blind Study of the Efficacy of Steroid Supplementation After Temporomandibular Joint Arthrocentesis
Brief Title: Efficacy of Steroid Supplementation After TMJ Rinsing for Pain Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201600060
Record Dates: First submitted 2013-01-11; First posted 2013-01-18 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Pain
Keywords: facial pain; temporomandibular joint; arthrocentesis; steroid
MeSH Terms: conditions — Pain; Facial Pain | interventions — Ringer's Lactate; triamcinolone hexacetonide; Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactated Ringers (Placebo Comparator): 1 cc of Lactated Ringers solution injected once after the TMJ rinsing procedure.
  Interventions: Drug: Lactated Ringers
- Triamcinolone acetonide (Active Comparator): 1 cc of triamcinolone acetonide (20 mg) injected once after the TMJ rinsing procedure.
  Interventions: Drug: Triamcinolone hexacetonide

INTERVENTIONS:
Drug: Lactated Ringers — Solution used for TMJ arthrocentesis procedure. 1 cc of Lactated Ringers solution injected once after the TMJ rinsing procedure.
  Arms: Lactated Ringers
Drug: Triamcinolone hexacetonide — 1 cc of triamcinolone hexacetonide (5 mg) injected once after the TMJ rinsing procedure.
  Other Names: Aristospan; steroid
  Arms: Triamcinolone acetonide

SUMMARY:
The hypothesis to be tested is temporomandibular joint (TMJ) rinsing followed by steroid injection is more efficacious than a placebo injection based on standard pain and physical measures that are recorded before and after treatment.

All procedures will be the same as if following normal TMJ arthrocentesis (rinsing) clinical care except that the patient will be randomly assigned to one of two groups: (1) TMJ rinsing followed by the injection of 1 cc (about ¼ of a teaspoon) of the same rinsing solution (this is the placebo) into the jaw joint; or (2) TMJ rinsing followed by the injection of 1 cc (about ¼ teaspoon) of a steroid (5 mg of triamcinolone hexacetonide) into the jaw joint. A pregnancy test (urine test) will be conducted on all women of child-bearing age to verify that the patient is not pregnant before the rinsing procedure. The patient will fill out a short questionnaire and have a short exam of the TMJ and jaw muscles at each appointment.

DETAILED DESCRIPTION:
Temporomandibular joint disorders are common and poorly understood in terms of etiology and pathogenesis. These disorders are multifactorial in origin including physical and psychosocial aspects; however, there is little understanding as to how much each of these components are associated with a particular diagnosis and subsequent treatment outcome of temporomandibular joint disorders. There is also a paucity of information regarding the relative effectiveness of different therapies for the treatment of patients with temporomandibular joint disorders. The identification of the least invasive and most efficacious therapy is vital to proper management of these patients with temporomandibular joint pain.

Patients enrolled into the study will be examined and treated at the Department of Oral and Maxillofacial Surgery. At the first appointment, they will be examined following standard procedures to determine if they would potentially benefit from the TMJ arthrocentesis procedure. If the patient meets the inclusion criteria for the study and with their informed consent, they will be required to complete a questionnaire about their physical and pain symptoms and undergo a standardized clinical exam. At the next appointment, the patients will undergo the standard clinical protocol for TMJ arthrocentesis with either only normal saline or normal saline with adjunctive steroids (triamcinolone hexacetonide). Follow-up appointments will be at 2 weeks, 6 weeks and 12 weeks where the pain VAS and clinical exams will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-80 years of age
* TMJ arthralgia
* Masticatory myalgia
* TMJ sounds
* History of at least 6 weeks use of occlusal appliance therapy

Exclusion Criteria:

* Contraindication to sedation including pregnancy or medical history
* History of previous TMJ procedure including arthrocentesis, arthroscopy or arthrotomy
* History of steroidal injection into TMJ
* History of trauma to TMJ
* TMJ pain longer than 3 years
* History of narcotic drug use on a scheduled basis
* Current active infection

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles G. Widmer, DDS, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Dentistry, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2013-2018 from facial pain referrals to the Oral and Maxillofacial Surgery Clinic.
Groups:
- Triamcinolone Acetonide: 1 cc of triamcinolone acetonide (20 mg) injected once after the TMJ rinsing procedure.
  Triamcinolone acetonide: 1 cc of triamcinolone acetonide (20 mg) injected once after the TMJ rinsing procedure.
Period: Overall Study
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactated Ringers | Triamcinolone Acetonide | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (17.5) | 52.7 (18.1) | 48.0 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Temporomandibular Joint Loading Pain [Median (Full Range); unit: units on a scale] — Loading pain is elicited by biting on a tongue blade on the opposite side of the temporomandibular joint that is tested. An ordinal scale pain rating is used that has a range of 0-3 with 0 representing "no pain" and 3 representing "severe pain".
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-Treatment in TMJ Loading Pain Rating at 12 Weeks
Description: TMJ loading pain is evaluated using ordinal scale ratings of 0-3 (none, mild, moderate, severe pain intensity).
Time Frame: Baseline and 12 weeks post-treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -1 [-2 to 0] | -2 [-3 to 0]

2. Secondary Outcome: Change From Pre-Treatment in TMJ Loading Pain Rating at 2 Weeks
Description: TMJ loading pain is evaluated using ordinal scale ratings of 0-3 (none, mild, moderate, severe pain intensity).
Time Frame: Baseline and 2 weeks post-treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -1 [-3 to 0] | -2 [-3 to 0]

3. Secondary Outcome: Change From Pre-Treatment in TMJ Loading Pain Rating at 6 Weeks
Description: TMJ loading pain is evaluated using ordinal scale ratings of 0-3 (none, mild, moderate, severe pain intensity).
Time Frame: Baseline and 6 weeks post-treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -1 [-2 to 2] | -2 [-3 to -1]

4. Secondary Outcome: Change From Pre-Treatment in Mandibular Range of Motion Without Pain at 2 Weeks
Description: Mandibular range of motion is measured in millimeters (mm) of vertical opening between the upper and lower central incisors plus vertical overlap of the incisors. These measures are made for jaw unassisted opening without pain, maximum unassisted opening and maximum assisted opening. Horizontal mandibular range of motion is measured in millimeters (mm) assessed for maximal right and left mandibular lateral movements and mandibular protrusion. A positive value represents an improvement (or larger range of motion) in mandibular opening/lateral movement.
Time Frame: Baseline and 2 weeks post-treatment
Measure: Mean (Standard Error); unit: mm
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
mm | 3.9 (2.4) | 9.7 (2.6)

5. Secondary Outcome: Change From Pre-Treatment in Mandibular Range of Motion at 6 Weeks
Description: as for outcome 4
Time Frame: Baseline and 6 weeks post-treatment
Measure: Mean (Standard Error); unit: mm
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
mm | 6.9 (2.8) | 7.4 (2.9)

6. Secondary Outcome: Change From Pre-Treatment in Mandibular Range of Pain-Free Motion at 12 Weeks
Description: as for outcome 4
Time Frame: Baseline and 12 weeks post-treatment
Measure: Mean (Standard Error); unit: mm
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
mm | 5.3 (2.1) | 10.0 (3.3)

7. Secondary Outcome: Change From Pre-Treatment Palpable Muscle Tenderness at 2 Weeks
Description: Palpable muscle tenderness of masticatory muscles using ordinal ratings of 0-3 (none, mild, moderate, severe pain to palpation) are summed. A standardized muscle palpation pressure is used at specific locations on each side of the face for a total of 20 locations. The range of possible scores is 0-60. The rating of each muscle palpation site is added for a composite muscle tenderness score.
Time Frame: Baseline and 2 weeks post-treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -2 [-16 to 7] | -1 [-5 to 2]

8. Secondary Outcome: Change From Pre-Treatment Palpable Muscle Tenderness at 6 Weeks
Description: as for outcome 7
Time Frame: Baseline and 6 weeks post-treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -1 [-16 to 3] | -1 [-5 to 2]

9. Secondary Outcome: Change From Pre-Treatment Palpable Muscle Tenderness at 12 Weeks
Description: as for outcome 7
Time Frame: Baseline and 12 weeks post-treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | 0 [-16 to 5] | -2 [-5 to 3]

10. Secondary Outcome: Number of Participants With Change From Pre-Treatment Joint Sounds in 2 Weeks
Description: Opening and closing sounds (click, course crepitus, fine crepitus) detected by palpation on left, right or both sides of face.
Time Frame: Baseline and 2 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
Participants | 1 | 5

11. Secondary Outcome: Number of Participants With Change From Pre-Treatment Joint Sounds in 6 Weeks
Description: as for outcome 10
Time Frame: Baseline and 6 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
Participants | 3 | 6

12. Secondary Outcome: Number of Participants With Change From Pre-Treatment Joint Sounds in 12 Weeks
Description: as for outcome 10
Time Frame: Baseline and 12 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
Participants | 4 | 5

13. Secondary Outcome: Change From Pre-Treatment Functional Pain (Chewing) at 2 Weeks
Description: Pain is assessed for average chewing pain intensity using a 100 mm visual analog scale with 0 representing "no pain" and 100 representing "the most intense chewing pain imaginable".
Time Frame: Baseline and 2 weeks post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -30 (6.1) | -37 (7.3)

14. Secondary Outcome: Change From Pre-Treatment Functional Pain (Chewing) at 6 Weeks
Description: as for outcome 13
Time Frame: Baseline and 6 weeks post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -33 (7.8) | -47 (9.2)

15. Secondary Outcome: Change From Pre-Treatment Functional Pain (Chewing) at 12 Weeks
Description: as for outcome 13
Time Frame: Baseline and 12 weeks post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
Number analyzed (Participants) | 10 | 12
units on a scale | -26 (9.6) | -43 (8.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Lactated Ringers | Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT01770912/Prot_SAP_000.pdf